CLINICAL TRIAL: NCT00636688
Title: Effect of Lifestyle Changes on Erectile Dysfunction in Obese Men: a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Dario Giugliano, MD,PhD, Department of Geriatrics and Metabolic Diseases, SUN Naples, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/2000
Record Dates: First submitted 2008-02-26; First posted 2008-03-14 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-03

CONDITIONS: Erectile Dysfunction
Keywords: Obesity; Lifestyle changes
MeSH Terms: conditions — Erectile Dysfunction; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Behavioral (Lifestyle Counseling)
  Interventions: Behavioral: Lifestyle - detailed advice
- 2 (Active Comparator): Control group
  Interventions: Behavioral: Control - general information

INTERVENTIONS:
Behavioral: Lifestyle - detailed advice — Detailed advice about how to achieve a loss of 10% or more in their total body weight by reducing caloric intake and increasing their level of physical activity
  Arms: 1
Behavioral: Control - general information — General information about healthy food choices and exercise
  Arms: 2

SUMMARY:
Healthy lifestyle factors are associated with maintenance of erectile function in men. To determine the effect of weight loss and increased physical activity on erectile and endothelial functions in obese men.

Randomized, single-blind trial of 110 obese men without diabetes, hypertension, or hyperlipidemia, who had erectile dysfunction that was determined by having a score of 21 or less on the International Index of Erectile Function (IIEF).

The 55 men randomly assigned to the intervention group received detailed advice about how to achieve a loss of 10% or more in their total body weight by reducing caloric intake and increasing their level of physical activity. Men in the control group (n = 55) were given general information about healthy food choices and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Obese, sedentary (<1 hour per week of physical activity) men with erectile dysfunction (a IIEF score lower than 22)and no evidence of participation in diet reduction programs within the last 6 months

Exclusion Criteria:

* Diabetes mellitus or impaired glucose tolerance (plasma glucose levels of 140-200 mg/dL [7.8-11.1 mmol/L] 2 hours after a 75-g oral glucose load)
* Impaired renal function, including macroalbuminuria, pelvic trauma, prostatic disease, peripheral or autonomic neuropathy
* Hypertension (blood pressure >140/90 mm Hg)
* Cardiovascular disease
* Psychiatric problems
* Use of drugs or alcohol abuse (500 g of alcohol per week in the last year).

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2000-10; Primary Completion 2003-04 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
IIEF (International Index Erectile Function) | two years

SECONDARY OUTCOMES:
Endothelial function, Circulating inflammatory markers | two years

CONTACTS AND LOCATIONS:
Overall Officials: Dario Giugliano, MD,PhD, Study Director — Department of Geriatrics and Metabolic Diseases, SUN Naples, Italy

REFERENCES:
- [Background] Bacon CG, Mittleman MA, Kawachi I, Giovannucci E, Glasser DB, Rimm EB. Sexual function in men older than 50 years of age: results from the health professionals follow-up study. Ann Intern Med. 2003 Aug 5;139(3):161-8. doi: 10.7326/0003-4819-139-3-200308050-00005. PMID 12899583
- [Result] Esposito K, Giugliano F, Di Palo C, Giugliano G, Marfella R, D'Andrea F, D'Armiento M, Giugliano D. Effect of lifestyle changes on erectile dysfunction in obese men: a randomized controlled trial. JAMA. 2004 Jun 23;291(24):2978-84. doi: 10.1001/jama.291.24.2978. PMID 15213209